CLINICAL TRIAL: NCT04301661
Title: Cellular Pharmacology and Platelet Effects of Abacavir and Lamivudine Anabolites
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-2749
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: HIV-1-infection
Keywords: NRTI; platelet
MeSH Terms: interventions — Blood Specimen Collection; abacavir, lamivudine drug combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, PBMC, RBC, dried blood spot (DBS), platelets, neutrophils
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ABC/3TC Cohort: Persons on abacavir/lamivudine-containing therapy as part of their standard HIV care will continue to take their prescribed HIV medications.
  Participants will be on study for 4 weeks, and will participate in directly observed therapy for the 4 weeks leading up to a single blood draw.
  Interventions: Other: Blood collection; Drug: Abacavir/lamivudine
- TAF/FTC Cohort: Persons on tenofovir alafenamide/emtricitabine-containing therapy as part of their standard HIV care will continue to take their prescribed HIV medications.
  Participants will be on study for 4 weeks, and will participate in directly observed therapy for the 4 weeks leading up to a single blood draw.
  Interventions: Other: Blood collection; Drug: Tenofovir alafenamide/emtricitabine
- Switch Cohort: Persons switching from abacavir/lamivudine-containing therapy as part of their standard HIV care will change to their newly prescribed regimen.
  Participants will be on study for 3 weeks, and will have blood drawn at Days 0, 1, 3, 7, 10, 14, 18, and 21 following their switch.
  Interventions: Other: Blood collection; Drug: Switch

INTERVENTIONS:
Other: Blood collection — Blood will be collected from participants at defined time points during the study to measure drug levels and assess platelet activity.
Drug: Abacavir/lamivudine — Participants who are already taking abacavir/lamivudine as part of standard HIV care will continue taking their therapy.
  Groups: ABC/3TC Cohort
Drug: Tenofovir alafenamide/emtricitabine — Participants who are already taking tenofovir alafenamide/emtricitabine as part of standard HIV care will continue taking their therapy.
  Groups: TAF/FTC Cohort
Drug: Switch — Participants who are planning to switch from abacavir/lamivudine as part of standard HIV care will change therapy to per the discretion of their HIV provider.
  Groups: Switch Cohort

SUMMARY:
This study will evaluate the intracellular pharmacokinetics and platelet effects of abacavir (ABC), lamivudine (3TC), tenofovir alafenamide (TAF), and emtricitabine (FTC) in persons living with HIV that are receiving these medications as part of standard HIV care.

Participants remaining on ABC/3TC- or TAF/FTC-containing therapy will be on study for 4 weeks, and will have two visits: a screening visit and one short PK visit consisting of a single blood draw at week 4.

Participants switching from their ABC/3TC-containing therapy will be on study for 3 weeks, and will have nine visits: a screening visit and 8 short PK visits consisting of a single blood draw at Day 0, 1, 3, 7, 10, 14, 18, and 21.

DETAILED DESCRIPTION:
Abacavir and lamivudine are recommended antiretroviral medications used in the treatment of human immunodeficiency virus (HIV) infection in the United States and globally. Both agents are nucleos(t)ide reverse transcriptase inhibitors (NRTIs), which exert their antiviral activity following entry into target cells and phosphorylation by intracellular kinases to their active anabolites, carbovir-triphosphate (CBV-TP) and lamivudine-triphosphate (3TC-TP). There is limited knowledge regarding the pharmacokinetic (PK) disposition of abacavir and lamivudine anabolites in red blood cells (RBCs), neutrophils, and platelets. Abacavir has also been linked with prothrombotic activity and an increased risk of cardiovascular events in patients on this therapy, central theories of which point towards interference with purinergic signaling due to its structural similarity to endogenous adenosine and guanosine. These findings have not been replicated with other NRTI medications, such as tenofovir. This pilot study will characterize the pharmacokinetics (PK) of these medications in different cell types of persons living with HIV (PLWH) on these therapies as part of clinical care, and will examine endogenous nucleotide levels and metabolic profiles through the use of metabolomics in platelets specifically to better understand what changes might be happening within this cell type with the use of these medications.

ELIGIBILITY:
Inclusion Criteria:

ABC/3TC Cohort:

* On abacavir 600 mg/lamivudine 300 mg-containing regimen as part of their ART for at least 6 months prior to entry
* HIV-1 RNA <200 copies/mL at screening and within the previous 6 months

TAF/FTC Cohort:

* On tenofovir alafenamide 25 mg/emtricitabine 200 mg-containing regimen as part of standard care for at least 6 months prior to entry
* HIV-1 RNA <200 copies/mL at screening and within the previous 6 months

Switch Cohort:

- Switching from an abacavir/lamivudine-containing regimen (to any other ART regimen not containing ABC/3TC) as part of standard care as recommended by their HIV provider

Exclusion Criteria:

* eGFR <50 mL/min/1.73 m2
* Platelet count <100,000 cells/mm3
* Current or previous use (within 30 days) of anticoagulant or antiplatelet medications (e.g., aspirin, P2Y12 inhibitors, vitamin K antagonists, anti-Xa inhibitors, thrombin inhibitors, etc.)
* History of cardiovascular event(s) (e.g., myocardial infarction, cerebrovascular accident (stroke), peripheral arterial thrombosis, etc.), platelet or bleeding disorders
* Pregnant or planning pregnancy
* Any uncontrolled medical, social, or mental-health issue(s) that, in the opinion of the investigators, could interfere with study participation or the study outcomes
* Inability to comply with directly observed dosing (i.e., lack of availability or ability to use video streaming technology)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons living with HIV receiving either abacavir/lamivudine or tenofovir alafenamide/emtricitabine as part of standard HIV care, or planning a switch from an abacavir/lamivudine-containing regimen.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Intracellular steady-state concentrations of abacavir and lamivudine anabolites in RBCs (also measured in DBS), PBMCs, platelets, and neutrophils. | (Week 4 in ABC/3TC and TAF/FTC Cohorts)
  Based on drug concentrations measured at week 4
Intracellular half-lives of abacavir and lamivudine anabolites in RBCs (also measured in DBS), PBMCs, platelets, and neutrophils. | (Days 0, 1, 3, 7, 10, 14, 18, 21 in Switch Cohort)
  Based on decline in drug concentrations between days 0 and 21.

OTHER OUTCOMES:
Intracellular concentrations of endogenous nucleotides measured in platelets from patients on abacavir- or tenofovir-containing therapy. | (Week 4 in ABC/3TC and TAF/FTC Cohorts; Days 0 and 21 in Switch Cohort)
Intracellular endogenous metabolites measured in platelets from patients on abacavir- or tenofovir-containing therapy. | (Week 4 in ABC/3TC and TAF/FTC Cohorts; Days 0 and 21 in Switch Cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Brooks, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No